CLINICAL TRIAL: NCT06448208
Title: Definition of PET REsponSe CrItEria for Neuroendocrine Tumors (PRESCIENT)
Brief Title: Defining Response Criteria for PET Scans for People With Neuroendocrine Tumors
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NeuroEndocrine Tumor Research Foundation (NETRF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24-100
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors
Keywords: PET scan; CT scan; 24-100
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People With Neuroendocrine Tumors having a PET/CT or MRI: This is a non-interventional observational study of imaging.
  Interventions: Diagnostic Test: positron emission tomography (PET) scans

INTERVENTIONS:
Diagnostic Test: positron emission tomography (PET) scans — Before and after treatment.

SUMMARY:
People with neuroendocrine cancer typically have imaging scans before and after treatment, including positron emission tomography (PET) scans. The scans are analyzed using a set of criteria that describes how the disease has responded to treatment. The purpose of this study is to establish new criteria for doctors to use when evaluating these PET scans. Researchers are testing whether these new criteria are useful for predicting whether a person's cancer gets better, gets worse, or stays the same. Researchers will also compare these new criteria to the current standard criteria for evaluating imaging scans.

ELIGIBILITY:
Subjects affected by histologically proven, somatostatin-receptor positive, metastatic or inoperable well-differentiated G1, G2 or G3 neuroendocrine tumors (NETs) candidate to receive PRRT with 177Lu-DOTATATE per standard of care.

Inclusion Criteria:

1. Histologically proven or cytologically confirmed, metastatic or inoperable NETs
2. Measurable disease as defined by RECIST 1.1.
3. Overexpression of somatostatin receptors of the target lesions at somatostatin receptor imaging (68Ga-DOTATATE or 64Cu-DOTATATE PET/CT) with SUV of lesions greater than normal liver at least in 1 metastasis.

Exclusion Criteria:

1. Neuroendocrine Carcinoma), small and large cell type; MIxed Neuroendocrine-Nonneuroendocrine Neoplasm (MiNEN).
2. Presence of somatostatin receptor negative lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering (MSK).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
validate the PRESCIENT criteria | 1 year
  On this prospective validation cohort, the prognostic value of each criteria for the 1-year PFS will be assessed, using a Cox regression model (stratified on the site) and the area under the receiver operating curve (AUC) for time-dependent outcome using inverse probability of censoring weighting.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bodei, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm